CLINICAL TRIAL: NCT03268187
Title: Biofeedback-based Relaxation Training or Self-alert Training to Alleviate Fatigue in Multiple Sclerosis Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rehazentrum Wilhelmshaven (Other)
Responsible Party: Principal Investigator, Carina Sander, Psychologist, Rehazentrum Wilhelmshaven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 009/2017
Record Dates: First submitted 2017-08-29; First posted 2017-08-31 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Fatigue; Multiple Sclerosis
Keywords: Cognitive Fatigue; Multiple Sclerosis; Biofeedback; Self-Alert Training; Vigilance; Autonomic potentials
MeSH Terms: conditions — Fatigue; Multiple Sclerosis | interventions — Biofeedback, Psychology; Relaxation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Alert Training (Experimental): Biofeedback-based Self-Alert Training Vigilance Task Questionnaires accessing apathy, fatigue, depression, sleep quality, sleep behavior
  Interventions: Device: Biofeedback; Behavioral: Self-Alert Training
- Relaxation Training (Active Comparator): Biofeedback-based Relaxation Training Vigilance Task Questionnaires accessing apathy, fatigue, depression, sleep quality, sleep behavior
  Interventions: Device: Biofeedback; Behavioral: Relaxation Training

INTERVENTIONS:
Device: Biofeedback — The skin conductance of the patient is measured and fed back to the patient via screen.
Behavioral: Self-Alert Training — Self-Alert Training
  Arms: Self-Alert Training
Behavioral: Relaxation Training — Relaxation Training
  Arms: Relaxation Training

SUMMARY:
The presented study compares the effectiveness of a biofeedback-based relaxation training with the effectiveness of a biofeedback-based self-alert training on the reduction of fatigue in multiple sclerosis patients using a between groups design. Furthermore, the relation of fatigue in multiple sclerosis patients and autonomic potentials as well as the performance in a vigilance task will be examined.

The relaxation training is based on the principle of progressive muscle relaxation according to Jacobsen. The patient is asked to tense all muscles in their face and perceive consciously the relaxation afterwards according to verbal cues. In the self-alert training condition, the patient will hear verbal cues to increase their attention. In both conditions the external cues given will be reduced in four phases until the patient has to cue himself. The patient is advised to track the changes in the skin resistance mirrored by biofeedback on a screen.

In both conditions the training will be split on two days. During the whole examination heart rate and skin resistance will be recorded. The allocation to the training happens randomly. On the first day the patient will complete questionnaires to survey depression and apathy and do a baseline vigilance task. Before and after the vigilance task the current fatigue status will be assessed using a visual analogue scale. Afterwards an introduction in the treatment method will be given.

On the second day the introduction into the training will be repeated. Afterwards a short time vigilance task will be done and questionnaires to survey fatigue and sleep behaviour and quality will be completed. Subsequently the last part of the training (no external cues) will be done. The examination will be completed by a long-time vigilance task. Before and after the vigilance task the current fatigue status will be assessed using a visual analogue scale.

It is hypothesised that especially the biofeedback-based self-alert training has a positive effect on fatigue and the vigilance performance in multiple sclerosis patients, as it increases the ectodermal activity and increases the sympathetic activation. It was shown that phasic changes of the skin resistance are correlated with an increase of neuronal activity in the brain areas relevant for vigilance (Critchley et al., 2002; Nagai et al., 2004). The relaxation training will reduce the sympatho-adrenergic excitation disposition and reduce the level of activity. Consequently, we do not expect an alleviation of the perceived fatigue according to our underlying model (Hanken et al., 2016). In addition, it is hypothesized that, independent from the treatment, autonomic potentials correlate with fatigue.

ELIGIBILITY:
Inclusion Criteria:

* at least a moderate cognitive fatigue (Fatigue Scale for Motor and Cognition minimum 22)
* clinical diagnosis of Multiple Sclerosis

Exclusion Criteria:

* psychiatric conditions independent from Multiple Sclerosis
* Pregnancy
* regular intake of psychostimulants
* no relapse in the last four weeks before
* no cortisone therapy in the last four weeks before
* patients with schizophrenia or serious personality disorders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2018-06-09 (Actual); Study Completion 2018-10-18 (Actual)

PRIMARY OUTCOMES:
Reaction Time of Vigilance Task (TAP) | Vigilance is measured at the beginning of the first day before the training introduction as well as after the training at the second day.
  Changes of the reaction time in the vigilance task
Subjective Fatigue (VAS) | Before and after the long-term vigilance tasks at day 1 and 2
  The current perceived fatigue

SECONDARY OUTCOMES:
Omissions and errors of Vigilance Task (TAP) | At day one before the introduction in the training and at day two after the training.
  The number of omissions and errors made in the Vigilance Task

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Hildebrandt, Prof, Study Director — Carl- von Ossietzky University Oldenburg
Locations (1):
- Rehazentrum Wilhelmshaven, Wilhelmshaven, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sander C, Braun N, Modes F, Schlake HP, Eling P, Hildebrandt H. Can biofeedback-based training alleviate fatigue and vigilance performance in fatigued MS patients? Neuropsychol Rehabil. 2022 Jan;32(1):131-147. doi: 10.1080/09602011.2020.1808023. Epub 2020 Aug 27. PMID 32851896